CLINICAL TRIAL: NCT02985177
Title: A Randomized Controlled Trial of a Combination of Analgesics for Pain Management in Children With a Suspected Fracture at Triage (CAST Trial)
Brief Title: A RCT of a Combination of Analgesics for Pain Management in Children With a Suspected Fracture
Acronym: CAST
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: We couldn't obtain funds for this study
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Sylvie Le May, Principal Investigator, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 99
Record Dates: First submitted 2016-10-25; First posted 2016-12-07 (Estimated); Last update posted 2022-11-23 (Actual); Status verified 2022-10

CONDITIONS: Emergency Service, Hospital; Child/Adolescent Problem; Acute Pain; Fentanyl; Ibuprofen; Analgesics, Opioid; Anti-inflammatory Agents, Non-steroidal
Keywords: Children; Musculoskeletal injury; Emergency department; Analgesia; Opioids
MeSH Terms: conditions — Emergencies; Acute Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- INF2.0 + IBU (Experimental): The participant will receive a dose of intranasal fentanyl (2.0 mcg/kg) AND a dose of oral ibuprofen (10 mg/kg).
  Interventions: Drug: INF2.0 + IBU
- INF1.0 + IBU (Active Comparator): The participant will receive a dose of intranasal (1.0 mcg/kg) AND a dose of oral ibuprofen (10 mg/kg).
  Interventions: Drug: INF1.0 + IBU

INTERVENTIONS:
Drug: INF2.0 + IBU — Analgesics
  Arms: INF2.0 + IBU
Drug: INF1.0 + IBU — Analgesics
  Arms: INF1.0 + IBU

SUMMARY:
MSK-I is the most common cause for ED visits for children with pain, with a child's risk of sustaining a fracture ranging from 27-42% by the age of 16 years. MSK-I is known to generate moderate to severe pain in most children and the ED serves as the critical entry point for these injured children. This study aims to provide rapid and sustained pain management for children presenting with a MSK-I in the ED. The investigators will compare the efficacy of two possible medication combinations of fentanyl intranasal (1.0 mcg/kg) + oral ibuprofen (10 mg/kg) and fentanyl intranasal (2.0 mcg/kg) + oral ibuprofen (10 mg/kg) for the rapid, adequate and sustained pain management of children with suspected fracture.

The investigators believe that the combination of different dosage of intranasal fentanyl with ibuprofen will lead to better pain treatment by providing a consistent and adequate level of analgesia throughout the entire ED visit, including prior to physician exam and during painful radiologic procedures.

DETAILED DESCRIPTION:
Pain management for children with a suspected fracture is suboptimal in the Emergency Department (ED). This type of musculoskeletal injury (MSK-I) often generates moderate to severe pain (> 49 mm on 0 to 100 mm Visual Analogue Scale (VAS)), and requires rapid and sustained pain management for the duration of the physical examination, diagnostic imaging (X-Ray), immobilization and occasionally fracture reduction. Current standard care includes the use of oral ibuprofen (IBU), a non-steroidal anti-inflammatory drug (NSAID), for mild-to-moderate MSK-I pain in the ED. However, ibuprofen has been shown to be inadequate for moderate-to-severe pain when used alone. A number of small/single centre studies suggest that intranasal fentanyl (INF) is effective for rapidly decreasing MSK-I related pain in children with a quick onset of 10 minutes and a peak action of 20 minutes. However, the duration of its analgesic effect is limited to a maximum of 60 minutes, which does not provide an optimal pain management for the duration of the ED stay, which typically lasts up to three hours. Typically, patients with a fracture have sustained pain throughout their ED stay due to imaging, splinting and repeated physical exams. Our objective is to examine the efficacy of a combination of intranasal and oral analgesics for pain management in children presenting to the ED with a suspected fracture. Our primary research question: For children presenting to the ED with a suspected fracture, is a combination of INF1.0 (1.0 mcg/kg, maximum dose of 100 mcg) and IBU (10 mg/kg, maximum dose of 600 mg) more efficacious than a combination of INF2.0 (2.0 mcg/kg, maximum dose of 100 mcg) and oral ibuprofen (10 mg/kg, maximum dose of 600 mg) to decrease pain at 15 minutes post-administration? Our primary hypothesis is: A combination of INF2.0 and IBU will be more efficacious than a combination of INF1.0 and IBU to decrease pain at 15 minutes post-administration.

Methods. Design: This study is a single-blind, two-arm, three-centre RCT of a combination of analgesics for pain management of children presenting to the ED with a suspected fracture will be performed. Settings: Children will be recruited in the following EDs: CHU Sainte-Justine (Montreal, QC), Stollery Children's Hospital (Edmonton, AB), and Children's Hospital of the London Health Sciences Centre (London, ON). Sample. Inclusion criteria: Will be include children: (a) with a pain score >49 mm on VAS at triage, (b) between the ages of 7 and 17 years, (c) presenting to the ED with a suspected fracture of the upper or lower limb, and (d) who can communicate in either French or English. Exclusion criteria: Will be exclude children with (a) known allergy to fentanyl or ibuprofen, (b) triage nurse suspicion of child abuse, (c) inability to self-report pain, (d) chronic pain that necessitates daily analgesic use, (e) NSAID or opioid analgesic use within the three hours prior to ED presentation, (f) trauma to >1 limb, (g) known hepatic or renal disease/dysfunction, (h) known bleeding disorder, (i) neuro-cognitive disability that precludes assent and/or participating in the study, (j) known history of obstructive sleep apnea (k) a suspected fracture of the nose, or (l) significant head injury, as determined by the clinical team/triage nurse.

Allocation and Randomization: A biostatistician, independent to our study team, will generate the randomization scheme that will consist of a computer-generated random listing of the treatment using a 1:1 allocation scheme. Randomization will be stratified by center using block-randomization (with permuted block sizes). Enrolled children will be allocated to (a) INF 1.0 mcg/kg (up to a maximum of 100 mcg) via intranasal atomization + oral IBU 10 mg/kg (up to a maximum of 600 mg) OR (b) INF 2.0 mcg/kg (up to a maximum of 100 mcg) via intranasal atomization + oral IBU 10 mg/kg (up to a maximum of 600 mg.

Sample Size: Accounting for a 10% attrition rate, we determined that enrollment of 172 participants would provide at least 90 % power to detect a 10 mm absolute difference in mean pain scores between groups at 15 minutes post-medication administration (T-15), at an alpha level of 5 %.

Primary efficacy outcome: Mean difference in pain scores between groups at 15 minutes post-medication administration (T-15) using the Visual Analogue Scale (VAS). Secondary outcomes: (a) Mean differences in pain scores between groups at 30 min (T-30), 60 min (T-60), 90 min (T-90), 120 min (T-120) after medication administration, during the medical examination (T-ME), and during radiographic procedure (T-XR), (b) the proportion of children administered a rescue analgesic in the 60 minutes following administration of study medication, (c) the proportion of children with adverse events at T-15, T-30, T-60, T-90, T-120, T-ME and T-XR, (d) the proportion of children with serious adverse events at T-15, T-30, T-60, T-90, T-120, T-ME and T-XR, (e) the proportion of children in each group with an RSS score > 3 (f) satisfaction of children and parents regarding pain management (T-120).

Relevance: In response to the persistent problem of inadequate and delayed analgesia, the investigators believe that a combination of rapidly acting (INF) and longer-acting (oral ibuprofen) medications will address both the delay in the time to effective analgesia and overall under-treatment of suspected fracture pain. The team anticipate that an RCT demonstrating the efficacy of a combination of fast and long-acting analgesics will significantly improve the treatment for children with a suspected fracture in the ED. The investigators hypothesize that use of INF2.0 and oral IBU will provide rapid pain relief that is sustained for the duration of the ED visit. Promotion of adequate acute pain treatment of children presenting to the ED will prevent the known short and long-term effects of inadequately treated pain in children previously demonstrated by our team, including unpleasant memories, stress and anxiety upon future visits to healthcare and compromised functional outcomes such as missed school.

ELIGIBILITY:
Inclusion Criteria:

* pain score >49 mm on the VAS at triage
* between the ages of 7 and 17 years
* presenting to the ED with a suspected fracture of the upper of lower limb
* who can communicate in either French or English

Exclusion Criteria:

* known allergy to fentanyl, ibuprofen
* triage nurse suspicion of child abuse
* inability to self-report pain
* chronic pain that necessitates daily analgesic use
* NSAID or opioid use within the three hours prior to ED presentation
* trauma to >1 limb
* known hepatic or renal disease/dysfunction
* known bleeding disorder
* neuro-cognitive disability that precludes assent and/or participating in the study
* known history of obstructive sleep apnea
* a suspected fracture of the nose
* significant head injury, as determined by the clinical team/triage nurse.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Mean difference in pain scores between groups | 15 minutes post-medication administration (T-15)
  Measure: Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
Mean difference in pain scores between groups | 30 min (T-30), 60 min (T-60), 90 min (T-90), 120 min (T-120) post-medication administration, during the medical examination (T-ME), and during radiographic procedure (T-XR)
  Measure: Visual Analogue Scale (VAS)
Proportion of children administered a rescue analgesic | Within 60 minutes following administration of study medication
  Measure: Clinical data (yes/no)
Proportion of children with adverse events in each group | 15 min (T-15), 30 min (T-30), 60 min (T-60), 90 min (T-90), 120 min (T-120) after medication administration, during the medical examination (T-ME), and during radiographic procedure (T-XR), 24 hours post-discharge from the ED
  At each assessment points, the research nurse will record the occurence of adverse events (clinical data)
Proportion of children with an RSS score > 3 in each group | 15 min (T-15), 30 min (T-30), 60 min (T-60), 90 min (T-90), 120 min (T-120) after medication administration, during the medical examination (T-ME), and during radiographic procedure (T-XR)
  At each assessment points, the research nurse will evaluate the child's sedation level using the Ramsay Sedation Scale (RSS)
Satisfaction of children and parents regarding pain management | 120 min (T-120) after medication administration
  Dichotomized question (yes/no)
Proportion of children with serious adverse events (SAE) in each group | After medication administration until discharge
  The research nurse will record the occurence of serious adverse events (clinical data)

CONTACTS AND LOCATIONS:
Overall Officials: Le May Sylvie, PhD, Principal Investigator — St. Justine's Hospital
Locations (3):
- Canada (3):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Children's Hospital London Health Sciences Centre, London, Ontario
  - CHU Sainte-Justine Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No